CLINICAL TRIAL: NCT00658060
Title: Exertional Muscle Fatigue In FMF Patients Evaluated By MRI And MR Spectroscopy Of The Thigh
Brief Title: Magnetic Resonance (MR) Spectroscopy In Familial Mediterranean Fever (FMF) Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Eshed Iris, MD, Sheba Medical Center
Other Study IDs: SHEBA-07-4632-IE-CTIL
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2008-04-14 (Estimated); Status verified 2008-04

CONDITIONS: Familial Mediterranean Fever
Keywords: FMF, Exertional leg pain
MeSH Terms: conditions — Familial Mediterranean Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: * 1.Fulfilling the Tel Hashomer criteria for the diagnosis of FMF [5].
  * 2.Suffering from episodes of exertional leg pain and or exertional ankle edema
  * 3.18-45 years old
  * 4.On a stable (≥ 2 weeks) dose of oral colchicine therapy
  * 5.Non-smokers
- 2: Control group
  * 1.Healthy subjects
  * 2.18-45 years old
  * 3.Non-smokers

SUMMARY:
Familial Mediterranean fever (FMF) is an inherited disorder of unknown etiology, characterized by recurrent episodes of fever, peritonitis and/or pleuritis.

Fever is the cardinal manifestation of FMF and is present in most attacks accompanied by abdominal pain.

Another clinical manifestation in patients with FMF is exertional muscle pain, usually in the thigh, which appears even after minor exercise or physical activity in young patients with generally good health (other than FMF) and in good physical condition. Some patients also complain of ankle edema after relatively minor physical activity, which subsides after a night rest. Although these manifestations are quite common in FMF patients and form part of the minor criteria for the diagnosis, the etiopathogenesis has not been examined.

The purpose of the suggested study is to evaluate and characterize the anatomical and biochemical changes in the muscles of the thigh and in the ankle triggered by physical activity in FMF patients complaining of exertional lower leg myalgias and edema after minor physical exercise.

ELIGIBILITY:
Inclusion Criteria:

1. Fulfilling the Tel Hashomer criteria for the diagnosis of FMF [5].
2. Suffering from episodes of exertional leg pain and or exertional ankle edema
3. 18-45 years old
4. On a stable (≥ 2 weeks) dose of oral colchicine therapy
5. Non-smokers

Exclusion Criteria:

1. with known peripheral vascular disease (PVD) and/or multiple risk factors for PVD (such as diabetes, hypertension, hyperlipidemia)
2. Suffering from muscular or neurological diseases not related to FMF
3. With elevated serum creatinine / liver enzymes/ creatine phosphokinase (CPK) levels.
4. Suffering from claustrophobia, or with metal fragments in body tissue, or with other contraindications for MRI.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with FMF, fulfilling the Tel Hashomer criteria for the diagnosis of FMF, suffering from episodes of exertional leg pain and or exertional ankle edema, 18-45 years old, on a stable (≥ 2 weeks) dose of oral colchicine therapy, Non-smokers
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2007-09

PRIMARY OUTCOMES:
change in spectroscopic appearance of muscle after exertion of muscle thigh | 1 hour

SECONDARY OUTCOMES:
change in muscle intensity signal after exertion | 1 hour
change in joint effusion status after exertion | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Iris Eshed, MD, Principal Investigator — Sheba Medical Center; Tammi Kushnir, PhD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Brik R, Shinawi M, Kasinetz L, Gershoni-Baruch R. The musculoskeletal manifestations of familial Mediterranean fever in children genetically diagnosed with the disease. Arthritis Rheum. 2001 Jun;44(6):1416-9. doi: 10.1002/1529-0131(200106)44:63.0.CO;2-6. PMID 11407703
- [Background] Bendahan D, Mattei JP, Guis S, Kozak-Ribbens G, Cozzone PJ. [Non-invasive investigation of muscle function using 31P magnetic resonance spectroscopy and 1H MR imaging]. Rev Neurol (Paris). 2006 Apr;162(4):467-84. doi: 10.1016/s0035-3787(06)75038-x. French. PMID 16585908